CLINICAL TRIAL: NCT06102837
Title: Preclinical and Clinical Research on Therapeutic Vaccines for Solid Tumors
Brief Title: Tumor Vaccines for Solid Tumors
Status: Recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Yu Yao, MD, Professor, Huashan Hospital
Other Study IDs: KY2023-846; 2022YFC3401605 (Other Grant/Funding Number: Grant from National Key R&D Program of China); 2022YFC3401600 (Other Grant/Funding Number: Grant from National Key R&D Program of China)
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Glioma; Solid Tumor
Keywords: Glioma; DC vaccine; Database; Biomarker; Artificial intelligence
MeSH Terms: conditions — Glioma | interventions — Cancer Vaccines; Radiotherapy; Drug Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- glioma patients receiving tumor vaccine
  Interventions: Biological: tumor vaccine; Radiation: Radiotherapy; Drug: Chemotherapy; Procedure: Surgery
- glioma patients receiving conventional treatment
  Interventions: Radiation: Radiotherapy; Drug: Chemotherapy; Procedure: Surgery
- non-tumor patients
  Interventions: Procedure: Surgery

INTERVENTIONS:
Biological: tumor vaccine — tumor vaccine produced by our team
  Groups: glioma patients receiving tumor vaccine
Radiation: Radiotherapy — conventional treatment in clincial
  Groups: glioma patients receiving conventional treatment; glioma patients receiving tumor vaccine
Drug: Chemotherapy — conventional treatment in clinical
  Groups: glioma patients receiving conventional treatment; glioma patients receiving tumor vaccine
Procedure: Surgery — conventional treatment in clinical

SUMMARY:
Glioma is the most common primary malignant intracranial tumor, characterized by limited clinical treatment options and extremely poor prognosis. There is an urgent need for the development of new technologies and clinical practice. With the advancement of immunotherapy, tumor therapeutic vaccines have emerged as a hot topic in the field of solid tumor immunotherapy. Several clinical trials have confirmed that tumor vaccines can improve the prognosis of glioma patients. Vaccines are the first systemic treatment technology in nearly 30 years that can simultaneously extend the overall survival of patients with newly diagnosed glioblastoma and recurrent glioblastoma in Phase III clinical trials. This novel approach holds significant clinical value and brings hope to large number of patients. Our team has previously developed a dendritic cell (DC) vaccine for glioma, and the phase II clinical trial has demonstrated that it can extend the prognosis of glioma patients. However, several patients benefit less from vaccine therapy. Therefore, the identification of molecular mechanisms that render patients unresponsive to vaccine treatment is critical to improving vaccine efficacy. This project aims to collect various types of clinical samples from patients, including glioma patients receiving tumor vaccine treatment, glioma patients receiving conventional clinical treatment without tumor vaccine, and non-tumor patients (hemorrhagic stroke, ischemic stroke, and traumatic brain injury). High-throughput sequencing techniques will be used to establish an immune microenvironment database, followed by bioinformatics analysis and molecular biology experiments to uncover the molecular mechanisms influencing vaccine efficacy. Artificial intelligence and deep learning technologies will be employed to extract molecular mechanisms related information from radiology images and pathology images. Ultimately, the project seeks to establish an integrated diagnostic and treatment model that combines imaging, pathology, and omics data to advance the clinical application of vaccines.

ELIGIBILITY:
Inclusion Criteria:

The patients with glioma patients/non-tumor patients (hemorrhagic stroke, ischemic stroke, and traumatic brain injury) in the Department of Neurosurgery of Huashan Hospital Affiliated to Fudan University who meet the following three conditions can be enrolled:

1. They were no age limit, male and female;
2. The pathological results of frozen section during operation were gliomas or non-tumor;
3. Tissue (6 mm * 6 mm) can be used for cell sorting on the basis of not affecting clinical routine diagnosis;
4. Sign informed consent.

Exclusion Criteria:

Patients who meet any of the following criteria will not be included in this study:

1. Participants in other clinical trials;
2. Pregnant women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing surgery at Huashan Hospital
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Transcriptomics | 48 months
  The issues collected will be used for transcriptome sequencing to measure gene expression level.
Immunomics | 48 months
  The issues collected will be used for TCR/BCR sequencing to measure clonality of lymphocytes
Proteomics | 48 months
  The issues collected will be used for proteomic sequencing to measure gene expression level in protein
Genomics | 48 months
  The issues collected will be used for whole genome sequencing or whole exome sequencing to measure gene mutations.
Radiomics | 48 months
  The features from images will be extracted using algorithm of Deep-learning or Radiomics
IHC analysis | 48 months
  Different expression level of proteins (CD3,CD8,B7-H4 et.al) in Gliomas with different grades and molecular subgroups will be measured using immunohistochemical.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China